CLINICAL TRIAL: NCT05415904
Title: Hantavirus Nephropathy in North-Eastern France : Severity Risk Factors and Prognostic Tools
Acronym: HANTA-NE
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, CORBEL Alice, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2022PI034
Record Dates: First submitted 2022-05-22; First posted 2022-06-13 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Hantavirus Nephropathy; Hantavirus Infection
Keywords: Acute kidney injury; Hantavirus infection; Hantavirus nephropathy
MeSH Terms: conditions — Hantavirus Infections; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HANTA-NE: All adult patient hospitalized for hantavirus infection between 01/01/2013 and 31/12/2022 in North Eastern France
  Interventions: Other: HANTA-NE

INTERVENTIONS:
Other: HANTA-NE — Observational cohort study

SUMMARY:
Hantaviruses are emerging pathogens responsible for hemorrhagic fever with renal syndrome. Severity risks factors aren't consensual in litterature, mostly related to scandinavian cohorts. A prognostic score was created to help patient's orientation in healthcare system but wasn't independantly validated (Hentzien, Emerging infectious diseases 2018).

This retrospective cohort of hantavirus infected hospitalized adults patients in the north-eastern quarter of France between 2013 and 2022 will specify the kidney damage during infection and risk factors for a severe form (defined par acute kidney injury KDIGO 3). The previous prognostic score performance will be evaluated in this cohort.

ELIGIBILITY:
Inclusion Criteria:

* hantavirus proven by serology infection
* age above 18 years
* Hospitalisation

Exclusion Criteria:

* age under 18 years
* fulfill opposition form

Ages: 18 Years to 125 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults patient hospitalized for hantavirus infection during study time frame.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Creatinin level | Through study completion, an average of 2 years
  Acute Kidney injury KDIGO 3
Hemorrhagic syndrome | Through study completion, an average of 2 years
  Major bleeding requiring blood transfusion
Death | Through study completion, an average of 2 years
  Death
Hospitalisation in intensive care unit | Through study completion, an average of 2 years
  Hospitalisation in intensive care unit

SECONDARY OUTCOMES:
Score performance to predict severity | Through study completion, an average of 2 years
  Correlation between severity predicted by the score and bio-clinical severity during hospitalization.
  Score composition :
  Hematuria = 7 Visual disorders = 8 Leucocyte count > 10 x 10^9 cells/L = 9 Nephrotoxic drug exposure (NSAID, iodinated contrast media, diuretics, renin angiotensin aldosterone system inhibitors, aminoglycosides, glycopeptides) = 10 Thrombocytopenia < or = 90 000/mm3 = 11
  Risk group according score scale 0-10 Low risk 11-19 intermediate risk 20-45 high risk
Hypotension | Through study completion, an average of 2 years
  Lowest systolic blood presure during hospitalisation < 90mmHg
Proteinuria | Through study completion,an average of 2 years
  Proteinuria during hospitalisation defined by proteinuria/creatininuria above 500 mg/g or equivalent
Urinary dipstick | Through study completion, an average of 2 years
  Leucocyturia or hematuria
ALAT, ASAT | Through study completion, an average of 2 years
  Liver cytolysis
calcium | Through study completion, an average of 2 years
  hypocalcemia, hypercalcemia
phosphorus | Through study completion, an average of 2 years
  hypophaspahtaemia, hyperphasphatemia
potassium | Through study completion, an average of 2 years
  hypokaliemia, hyperkaliemia
sodium | Through study completion, an average of 2 years
  blood sodium level disorders
bicarbonate blood level | Through study completion, an average of 2 years
  metabolic acidosis, metabolic alcalosis
Heamoglobin | Through study completion, an average of 2 years
  Anemia
platelets level | Through study completion, an average of 2 years
  thrombocytemia
Urine output | Through study completion, an average of 2 years
  Polyruria above 3 L/day

CONTACTS AND LOCATIONS:
Overall Officials: Alice CORBEL, M.D., Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Central Hospital, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided